CLINICAL TRIAL: NCT04606199
Title: Pilot Testing of an Ecological Momentary Mindfulness-based Intervention (EMMI) for People With Early Life Adversity
Brief Title: Examine the Effects of Meditation on Daily Psychological Stress Responses in Woman With a History of Child Adversity
Acronym: EMMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Harvard University (Other); National Institute on Aging (NIA) (NIH); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-27198; K99AG062778 (NIH)
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Stress; Psychological Stress; Child Maltreatment; Depressive Symptoms; Signs and Symptoms; Psychological Distress; Psychological
Keywords: Mindfulness; Adverse childhood experiences; Stress appraisals; Affect; Daily psychological stress responses; Stress; Depressive symptoms
MeSH Terms: conditions — Stress, Psychological; Depression; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: A Micro-Randomized Trial (MRT) is a design that randomly assigns an intervention at each notification time point (similar to a crossover design in that each participant is randomized to both conditions at different times, except in the MRT the crossover occurs at multiple times): Participants use the study app for 30 days and receive three notifications per day. At each notification time point, participants complete an Ecological Momentary Assessment (EMA) of their current psychological stress states (pre-EMA). Then, at each notification, each participant is randomized (50 percent probability) to either receive a mindfulness-based intervention or not. Thus, participants are randomized many times over the 30-day study. Approximately thirty minutes post-randomization, an EMA is obtained again to assess psychological stress states (post-EMA). A treatment effect is examined by comparing psychological stress responses after a mindfulness-based intervention compared to no intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Since the study uses a MRT design (each participant is randomized multiple times), the investigator and outcomes assessor do not know at what time points participants are assigned to an intervention or not over the course of this 30-day study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based intervention (Experimental): Participants will be randomly assigned to an app-based intervention that includes brief (<5 min) audio-guided mindfulness and compassion-based practices.
  Interventions: Behavioral: Mindfulness-based intervention, up to 5 minutes 0-3 times/day
- No intervention (No Intervention): Participants will continue their normal activities and not practice any form of mindfulness mediation at the time of app-notification.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention, up to 5 minutes 0-3 times/day — The intervention consist of mindfulness and compassion-based practices that are selected to maximize their effect on stress targets. Interventions include, for example, practices that focus on the breath/body (e.g., 3 minute breathing space; compassionate body scan; five senses mediation), on increasing participants' inner resources (e.g., imaging a safe person or safe place), on reducing negative affect (e.g., self-compassion and acceptance-based practices), or on increasing positive emotions (e.g., gratitude practice; metta practices).
  Arms: Mindfulness-based intervention

SUMMARY:
The aim of the Everyday Moments of Mindfulness (EMMI) study is to test whether brief mindfulness-based practices will improve daily psychological stress responses in women (age 30-60) who report a history of early life adversity. Following a baseline visit (remotely or in person), participants complete daily surveys and audio-guided mindfulness-based practices in everyday life via the study app. Specifically, participants receive app-notifications three times/day (morning, afternoon, evening) to complete daily surveys of current stressors and psychological states. At each notification, each participant is then randomly assigned to either receive a mindfulness-based intervention or not (max of 3 interventions/day). Thus, participants are randomized many times over the course of this 30-day study. At the end of the study, participants complete a follow-up visit (remotely or in person).

DETAILED DESCRIPTION:
The aim of the present study is to test whether brief app-based mindfulness and compassion practices will improve daily psychological stress responses in a sample of adult women (age 30-60) who report a history of early life adversity. The study will incorporate surveys and mindfulness-based intervention practices into everyday life using mobile technology (study app). Participants receive app-notifications three times/day (morning, afternoon, evening) to complete Ecological Momentary Assessments (EMAs) of current psychological stress states (pre-EMA; e.g., stress appraisals, affect, perseverative cognitions, self-criticism, social connection). At each notification, each participant is then randomized to either receive a mindfulness-based intervention (described in detail below) or no intervention. Thus, each participant is randomized many times over this 30-day study (Micro-Randomized Trial, MRT). Psychological stress states are again measured approximately 15 min post-randomization (post-EMA; e.g., stress appraisals, affect, perseverative cognitions, self-criticism, social connection) to assess a treatment effect by comparing psychological stress responses after a mindfulness-based intervention vs. no intervention. The MRT will continue for 30 days. All study participants will be asked to fill out questionnaires at baseline and post-intervention (after 30 days). Weekly measures of depressive symptoms are also obtained. A trained research assistant will monitor participant adherence and address potential difficulties.

Mindfulness-based intervention: The intervention consists of mindfulness and compassion-based practices. For example, practices focus on the breath/body (e.g., 3 minute breathing space; compassionate body scan; five senses mediation), on increasing participants' inner resources (e.g., imaging a safe person or safe place), on reducing negative affect (e.g., self-compassionate and acceptance-based practices), or on increasing positive emotions (e.g., gratitude practice; metta practices). All interventions are brief (≤5 minutes) and audio-guided.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* age 30-60
* reports at least two adverse childhood experiences on the 10-item Adverse Childhood Experiences (ACE) scale
* reports at least mild depressive symptoms (Patient Health Questionnaire ≥ 5)
* has access to a personal smartphone

Exclusion Criteria:

* Non-English speaker or unable to provide informed consent
* Current regular mindfulness practice (exclude if >20 min/week)
* Diagnosis of severe psychiatric disorders, including psychosis/schizophrenia, bipolar disorder, post-traumatic stress disorder (PTSD), alcohol/substance-use disorder, major depressive disorder (PHQ-9 ≥ 15), and self-harm or suicidal ideation (PHQ-9, item 9).
* Unstable medication use and psychotherapy treatment (<3 months).

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-representation of gender identity.
Enrollment: 53 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie E Mayer, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness-based Micro-intervention: Overview: The study used a micro-randomized trial design in which participants received app-notifications three times/day (morning, afternoon, evening). At each notification time-point, participants had a 50% chance of receiving either a mindfulness-based intervention or no intervention (described below). Thus, each participant was randomized many times over this 30-day study.
  Mindfulness-based intervention: Participants randomly assigned to an app-based mindfulness intervention were instructed to do a brief (<5 min) audio-guided mindfulness practice. The intervention was randomly selected out of 12 practices that consisted of mindfulness and compassion-based practices (e.g., 3 minute breathing space; compassionate body scan; five senses meditation, imagining a safe person or safe place, self-compassion and acceptance-based practices; gratitude practice; metta practices).
  No intervention: Participants randomly assigned to "no intervention" just continued their normal activities; they did not practice any form of mindfulness mediation at the time of app-notification.
Period: Overall Study
Arm/Group | Mindfulness-based Micro-intervention
Started | 53
Completed | 51
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mindfulness-based Micro-intervention
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.85 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 9
  White | 24
  More than one race | 4
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53
9-item Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The 9-item Patient Health Questionnaire (PHQ-9) has a total score scale range of 0 to 27, with higher values indicating more depressive symptoms.
  units on a scale | 8.62 (2.33)
7-item General Anxiety Disorder (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — The 7-item General Anxiety Disorder (GAD-7) questionnaire assesses symptoms of anxiety in the past 2 weeks. The total score scale ranges from 0 to 21, with higher values indicating higher anxiety.
  units on a scale | 9.75 (4.99)
10-item Perceived Stress Scale (PSS) [Mean (Standard Deviation); unit: units on a scale] — The 10-item Perceived Stress Scale (PSS) has a total score scale range of 0 to 40, with higher values indicating higher perceived stress.
  units on a scale | 23.47 (5.84)

OUTCOME MEASURES:

1. Primary Outcome: Change in Stressor Demands, as Measured by Ecological Momentary Assessment (EMA)
Description: Stressor demands were measured by computing a total mean score of "I feel stressed, anxious, overwhelmed" and "I feel strained, upset, overburdened." The total mean score ranges from 1 to 7, with higher scores indicating greater stressor demands. Stressor demands were assessed at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of stressor demands immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Change in stressor demands was calculated as post-EMA minus pre-EMA.
Time Frame: From pre-EMA (immediately prior to intervention randomization) to post-EMA, approximately 15 minutes post-randomization, over a period of 30 days.
Population: All 53 participants were included in the analysis. There was a total of 90 possible decision points per participant. Unimputed data are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Groups:
- Mindfulness-based Intervention: Participants were randomly assigned to an app-based intervention that included brief (<5 min) audio-guided mindfulness and compassion-based practices.
  Mindfulness-based intervention, up to 5 minutes 0-3 times/day: The intervention consisted of mindfulness and compassion-based practices that were selected to maximize their effect on stress targets. Interventions included, for example, practices that focused on the breath/body (e.g., 3 minute breathing space; compassionate body scan; five senses mediation), on increasing participants' inner resources (e.g., imaging a safe person or safe place), on reducing negative affect (e.g., self-compassion and acceptance-based practices), or on increasing positive emotions (e.g., gratitude practice; metta practices).
- No Intervention: Participants continued their normal activities and did not practice any form of mindfulness mediation at the time of app-notification.
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 1547 | 1653
score on a scale | -.0950 (.84983) | .0009 (.74960)

2. Primary Outcome: Change in Negative Affect, as Measured by Ecological Momentary Assessment (EMA)
Description: Negative affect was measured by computing a total mean score of "I feel sad, downhearted, unhappy" and "I feel angry, irritated, frustrated." The total mean score ranges from 1 to 7, with higher scores indicating greater negative affect. Negative affect was measured at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of negative affect immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Change in negative affect was calculated as post-EMA minus pre-EMA.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 1542 | 1650
score on a scale | -.0610 (.83630) | .0018 (.72844)

3. Secondary Outcome: Change in Coping Resources, as Measured by Ecological Momentary Assessment (EMA)
Description: Coping resources were measured by computing a total mean score of "I feel in control, coping well, on top of things" and "I feel capable, competent, managing well." The total mean score ranges from 1 to 7, with higher scores indicating greater coping resources. Coping resources were measured at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of coping resources immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Change in coping resources was calculated as post-EMA minus pre-EMA.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 1543 | 1651
score on a scale | .1134 (.90167) | .0112 (.76279)

4. Secondary Outcome: Change in Positive Affect, as Measured by Ecological Momentary Assessment (EMA)
Description: Positive affect was measured by computing a total mean score of "I feel joyful, glad, happy", "I feel calm, peaceful, quiet" and "I feel grateful, appreciative, thankful." The total mean score ranges from 1 to 7, with higher scores indicating greater positive affect. Positive affect was assessed at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of positive affect immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Changes in positive affect was calculated as post-EMA minus pre-EMA.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 1542 | 1648
score on a scale | .1288 (.82500) | .0038 (.66488)

5. Secondary Outcome: Change in Perseverative Cognitions, as Measured by Ecological Momentary Assessment (EMA)
Description: Perseverative cognitions were measured by computing a total mean score of "I feel worried, concerned, uneasy" and "I dwell, ruminate, brood on my personal problems and feelings." The total mean score ranges from 1 to 7, with higher scores indicating greater perseverative cognitions (greater rumination/worry). Perseverative cognitions were assessed at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of perseverative cognitions immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Change in perseverative cognitions was calculated as post-EMA minus pre-EMA.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 1540 | 1648
score on a scale | -.1088 (.78940) | -.0322 (.69380)

6. Secondary Outcome: Change in Self-criticism, as Measured by Ecological Momentary Assessment (EMA)
Description: Self-criticism were measured by computing a total mean score of "I feel self-critical, self-blaming, self-loathing" and "I feel inadequate, not good enough, unworthy." The total mean score ranges from 1 to 7, with higher scores indicating greater self-criticism. Self-criticism was assessed at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of self-criticism immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Change in self-criticism was calculated as post-EMA minus pre-EMA.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 1540 | 1647
score on a scale | -.0932 (.74596) | -.0188 (.64742)

7. Secondary Outcome: Change in Social Connection, as Measured by Ecological Momentary Assessment (EMA)
Description: Social connection was measured by computing a total mean score of "I feel love, closeness, trust" and "I feel lonely, isolated, disconnected" [reverse coded]). The total mean score ranges from 1 to 7, with higher scores indicating greater social connection. Social connection was assessed at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of social connection immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Change in social connection was calculated as post-EMA minus pre-EMA.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 1540 | 1647
score on a scale | .0880 (.77520) | -.0134 (.69068)

8. Secondary Outcome: Change in Contextualized Stressor Demands, as Measured by Ecological Momentary Assessment (EMA)
Description: Participants were asked about current stressors ("Is there a stressful situation in your day right now?") using a 7-point scale (1 = "not at all"; 7 = "extremely"). If a response other than "not at all" was endorsed, contextualized stressor demands ("How demanding is it to deal with this situation well right now?") was measured on a 7-point scale (1 = "not at all"; 7 = "extremely") at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of contextualized stressor demands immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Change in contextualized stressor demands was calculated as post-EMA minus pre-EMA.
Time Frame: as for outcome 1
Population: All 53 participants were included in the analysis. There was a total of 90 possible decision points per participant at which they were asked about current stressors ("Is there a stressful situation in your day right now?"). If a response other than "not at all" was endorsed, contextualized stressor demands were assessed. Unimputed data are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 823 | 870
score on a scale | -.0984 (1.15313) | -.0161 (1.08752)

9. Secondary Outcome: Change in Contextualized Coping Resources, as Measured by Ecological Momentary Assessment (EMA)
Description: Participants were asked about current stressors ("Is there a stressful situation in your day right now?") using a 7-point scale (1 = "not at all"; 7 = "extremely"). If a response other than "not at all" was endorsed, contextualized coping resources ("Do you feel like you can handle this situation well right now?") were measured on a 7-point scale (1 = "not at all"; 7 = "extremely") at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of contextualized coping resources immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Change in contextualized coping resources was calculated as post-EMA minus pre-EMA.
Time Frame: as for outcome 1
Population: All 53 participants were included in the analysis. There was a total of 90 possible decision points per participant at which they were asked about current stressors ("Is there a stressful situation in your day right now?"). If a response other than "not at all" was endorsed, contextualized coping resources were assessed. Unimputed data are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 823 | 870
score on a scale | .0668 (1.01529) | -.0172 (.85195)

10. Secondary Outcome: Change in Negative Stressor Impact, as Measured by Ecological Momentary Assessment (EMA)
Description: Participants were asked about current stressors ("Is there a stressful situation in your day right now?") using a 7-point scale (1 = "not at all"; 7 = "extremely"). If a response other than "not at all" was endorsed, negative stressor impact ["How much does this situation negatively impact you right now (e.g., interferes with your well-being or functioning)?"] was measured on a 7-point scale (1 = "not at all"; 7 = "extremely") at notification time points 3 times/day over a 30-day period. At each notification time point, participants completed EMAs of negative stressor impact immediately prior to intervention randomization (pre-EMA) and approximately 15 minutes post randomization (post-EMA). Change in negative stressor impact was calculated as post-EMA minus pre-EMA.
Time Frame: as for outcome 1
Population: All 53 participants were included in the analysis. There was a total of 90 possible decision points per participant at which they were asked about current stressors ("Is there a stressful situation in your day right now?"). If a response other than "not at all" was endorsed, negative stressor impact were assessed. Unimputed data are reported here.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Decision points
Arm/Group | Mindfulness-based Intervention | No Intervention
Number analyzed (Participants) | 53 | 53
Number analyzed (Decision points) | 823 | 870
score on a scale | -.1021 (1.13098) | -.0736 (1.02853)

11. Other Pre Specified Outcome: Change in Depressive Symptoms, as Measured by the 9-item Patient Health Questionnaire (PHQ-9).
Description: The 9-item Patient Health Questionnaire (PHQ-9) has a total score scale range of 0 to 27, with higher values indicating more depressive symptoms. Change in depressive symptoms was calculated as post-intervention minus baseline values.
Time Frame: Baseline to post-intervention, over a period of 30 days.
Population: Participants who completed both pre and post measures were included (n = 51).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Micro-intervention
Number analyzed (Participants) | 51
score on a scale | -2.61 (4.78)

12. Other Pre Specified Outcome: Change in Perceived Stress, as Measured by the 10-item Perceived Stress Scale (PSS)
Description: The 10-item Perceived Stress Scale (PSS) has a total score scale range of 0 to 40, with higher values indicating higher perceived stress. Change in perceived stress was calculated as post-intervention minus baseline values.
Time Frame: Baseline to post-intervention, over a period of 30 days.
Population: Participants who completed both pre and post measures were included (n = 51).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Micro-intervention
Number analyzed (Participants) | 51
score on a scale | -3.76 (5.55)

13. Other Pre Specified Outcome: Change in Anxiety, as Measured by the 7-item General Anxiety Disorder (GAD-7) Questionnaire
Description: The 7-item General Anxiety Disorder (GAD-7) questionnaire assesses symptoms of anxiety in the past 2 weeks. The total score scale ranges from 0 to 21, with higher values indicating higher anxiety. Change in anxiety was calculated as post-intervention minus baseline values.
Time Frame: Baseline to post-intervention, over a period of 30 days.
Population: Participants who completed both pre and post measures were included (n = 51).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-based Micro-intervention
Number analyzed (Participants) | 51
score on a scale | -2.14 (4.59)

ADVERSE EVENTS:
Time Frame: Baseline to post-intervention, an anticipated average of 30 days.
Arm/Group | Mindfulness-based Micro-intervention
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT04606199/Prot_SAP_000.pdf